CLINICAL TRIAL: NCT03735472
Title: National Observational Study of the Thoraflex™ Hybrid Vascular Prosthesis in the Replacement of the Aortic Arch and the Treatment of Aneurysm/dissection of the Descending Thoracic Aorta
Brief Title: Study of the Thoraflex™ Hybrid Device for the Treatment of Aneurysm/dissection of the Descending Thoracic Aorta
Status: Completed | Type: Observational
Sponsor: Vascutek Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: EPI-Flex
Record Dates: First submitted 2015-12-16; First posted 2018-11-08 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-11

CONDITIONS: Aortic Arch; Aneurysm, Dissecting
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (1):
- Aneurysm/Dissection: Thoraflex™ Hybrid
  Interventions: Device: Thoraflex™ Hybrid

INTERVENTIONS:
Device: Thoraflex™ Hybrid — The Thoraflex™ Hybrid device is particularly suited to the treatment of extended lesions of the ascending aorta, the aortic arch and the descending aorta, which constitute a major challenge in cardiovascular surgery.
  It enables, during a single surgical operation, combination of the "Frozen Elephant Trunk" technique and a 4-branch prosthesis of the aortic arch, thus enhancing the arsenal of the surgeon in the treatment of complex diseases of the aortic arch.

SUMMARY:
The purpose of this national observational study is to evaluate the Thoraflex™ Hybrid vascular prosthesis in the replacement of the aortic arch and the treatment of aneurysm/dissection of the descending thoracic aorta in relation to morbidity-mortality, visceral malperfusions, neurological and renal complications, endoleak and evolution of the aortic thoracic stent over time.

DETAILED DESCRIPTION:
Quality control will be performed continuously at various stages of the error correction process, according to the sponsor's Standard Operating Procedures.

Systematic coherence control procedures will be implemented and documented. The correction procedures will be tracked. For the study data, requests (Queries) will be issued and transmitted to the various centres for resolution.

To ensure data quality, a Monitoring Plan will be implemented. This plan will detail the frequency of visits or check-ups and the proportion of the data verified. It is expected that at least 10% of the data will be verified.

The monitoring factors in relation to the quality of electronic case report form completion will be performed by one of the Clinical Research Associates.

The participating physicians will be automatically contacted in the event of the absence of data entry after inclusion of patients and/or dates of scheduled visits and planned controls.

All of the analyses will be managed by the Direction de la Recherche Clinique et de l'Innovation of CHU Amiens. The statistical analysis software to be used is SAS (version 9.1). According to the target population, a sample of approximately 80 to 100 patients is anticipated, which would enable accuracy of ± 8.5 to 9.5% for an estimation of an event rate of around 25%.

During implementation of the study, the observers will be asked to minimise any missing data. The data collected is comparable to usual practice, which should be available from the original medical record. However, in the event of absence of the latter, the note missing data will be added to the data collection form. Several measures will be taken to avoid patients being lost to follow-up.

The study documents provided to the observers for initiation emphasise the fundamental importance of patient follow-up and the collection of data during the entire study. If necessary, scientific societies as well as the French National Authority of Health (HAS) may remind the observers of their obligation to actively participate in the existing national observational study.

The observer will obtain the means to contact the patient, his/her General Practitioner or close friend/next of kin.

Demographic and medical data of patients and follow-up descriptive data will be reflected in the patient population included.

Qualitative parameters are described by their frequency distribution and related bilateral 95% confidence intervals, quantitative parameters by their average, standard deviation minimum, maximum, median and quartiles, number of missing values.

Each of the rates corresponding to the study criteria is analysed by calculating the frequencies of distribution and related bilateral 95% confidence intervals (95% CI).

The rate of events over time will be described by a survival curve using the Kaplan Meier method and the related Kaplan Meier estimators will be calculated.

On an exploratory basis, the criteria in the study will also be analysed according to the basic characteristics of the patients:

* Age (in categories)
* Sex
* Indications.

ELIGIBILITY:
Inclusion Criteria:

• Patient presenting an aneurysm/dissection of the thoracic aorta of the aortic arch and/or the descending thoracic aorta, and necessitating a procedure of the "Elephant Trunk" type, with the Thoraflex™ Hybrid hybrid vascular prosthesis.

Exclusion Criteria:

* Patient having refused to sign the Consent form to the use of his/her data.
* Patient residing abroad, for whom follow-up is not possible.
* Patient with active endocarditis
* Patient who has received a post-infarction septal repair.
* A list of all of the patients who have received the Thoraflex™ Hybrid hybrid vascular prosthesis but not participating in the observational study will be documented, as well as the reasons for non-inclusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient presenting an aneurysm/dissection of the thoracic aorta of the aortic arch and/or the descending thoracic aorta and necessitating surgery of the Elephant Trunk type. To meet the requirements of the French National Authority for Health, this study will include all the patients treated with the Thoraflex™ Hybrid hybrid vascular prosthesis. Any surgeon practising in France and wishing to inplant a Thoraflex™ Hybrid hybrid vascular prosthesis will be available from the coordinating observer.
Sampling Method: Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2024-11 (Actual)

PRIMARY OUTCOMES:
Patients who did not die, nor suffered paraplegia due to the prosthesis, nor had complications linked to the procedure and surgical conversion | 30 days post-operative
  Percentage of patients who did not die, nor suffered paraplegia due to the prosthesis, nor had complications linked to the procedure and surgical conversion for 30 days post-operative

SECONDARY OUTCOMES:
Technical success | Within 30 days of intervention; Between 3 and 6 months; then documented by the patient's clinical course up to 3 years.
  is defined as the placement and deployment of the a Vascutek Thoraflex™ Hybrid Device in the absence of mortality, conversion to conventional open surgical repair, failed patency, evidence of an unanticipated distal type I or type III endoleak on pre-discharge CT scan
Death | Within 30 days of intervention; Between 3 and 6 months; then documented by the patient's clinical course up to 3 years.
  Death linked to the device, to the procedure, all causes
Transitory paraplegia/Para-paresis | Within 30 days of intervention; Between 3 and 6 months; then documented by the patient's clinical course up to 3 years.
  Transitory paraplegia/Para-paresis
Follow-up surgery | Within 30 days of intervention; Between 3 and 6 months; then documented by the patient's clinical course up to 3 years.
  Follow-up Surgery linked/not linked to the device
Complications linked to the device | Within 30 days of intervention; Between 3 and 6 months; then documented by the patient's clinical course up to 3 years.
  No plication, torsion, occlusion and thrombosis of the device, Leak-tightness of the polyester prosthesis, Change over time of the thoracic stent graft
Rates of visceral malperfusion, neurological, renal, cardiac, respiratory and Haemorrhagic complications | Within 30 days of intervention; Between 3 and 6 months; then documented by the patient's clinical course up to 3 years.
  Rates of visceral malperfusion, neurological, renal, cardiac, respiratory and Haemorrhagic complications

CONTACTS AND LOCATIONS:
Overall Officials: Professor Thierry Caus, Principal Investigator — Centre Hospitalier Universitaire. Heart, Chest and Vascular Centre, AMIENS
Locations (37):
- France (37):
  - Centre Hospitalier University (University Hospital centre), Amiens
  - CHU Angers, Angers
  - CH De La Region D Annecy, Annecy
  - CHU-Hopital Jean Minjoz, Besançon
  - Hopital Cardio-Vasculaire Louise Pradel, Bron
  - CHU Cote De Nacre, Caen
  - CHU - Hopital Gabriel Montpied, Clermont-Ferrand
  - CHU Hopital Henri Mondor, Créteil
  - CHU - Hopital Du Bocage, Dijon
  - CHU Hopital A. Michallon, Grenoble
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - CHRU Lille, Lille
  - Clinique De La Sauvegarde, Lyon
  - CHU Hopital La Timone, Marseille
  - Hopital Clinique Claude Bernard, Metz
  - Hopital De Mercy, Metz
  - CHU Hopital Arnaud De Villeneuve, Montpellier
  - CHU - Hopital Brabois, Nancy
  - CHU - Hopital Guillaume et Rene Laenec, Nantes
  - Hopital Prive Les Franciscaines, Nîmes
  - Groupe Hospitalier Pitié-Salpêtrière, Vascular Surgery Department, Paris
  - Groupe Hospitalier La Pitie Salpetriere, Paris
  - Hopital Bichat, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU - Hopital Haut Leveque, Pessac
  - CHU - Hopital Robert Debre, Reims
  - CHU - Hopital Pontchaillou, Rennes
  - CHU Charles Nicolle, Rouen
  - Centre Cardiologique Du Nord, Saint-Denis
  - CH Felix Guyon, Saint-Denis
  - CHU De Saint Etienne, Saint-Etienne
  - Hopitaux Universitaires - Nouvel Hopital Civil, Strasbourg
  - Hôpital Rangueil, Cardiothoracic Surgery Department, Toulouse
  - Clinique Pasteur, Toulouse
  - CHU De Tours, Tours
  - Clinique Du Tonkin - Medipole, Villeurbanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bortone AS, Schena S, D'Agostino D, Dialetto G, Paradiso V, Mannatrizio G, Fiore T, Cotrufo M, de Luca Tupputi Schinosa L. Immediate versus delayed endovascular treatment of post-traumatic aortic pseudoaneurysms and type B dissections: retrospective analysis and premises to the upcoming European trial. Circulation. 2002 Sep 24;106(12 Suppl 1):I234-40. PMID 12354739
- [Background] Arko FR, Lee WA, Hill BB, Olcott C 4th, Harris EJ, Dalman RL, Fogarty TJ, Zarins CK. Impact of endovascular repair on open aortic aneurysm surgical training. J Vasc Surg. 2001 Nov;34(5):885-91. doi: 10.1067/mva.2001.118816. PMID 11700491
- [Background] Karck M, Chavan A, Hagl C, Friedrich H, Galanski M, Haverich A. The frozen elephant trunk technique: a new treatment for thoracic aortic aneurysms. J Thorac Cardiovasc Surg. 2003 Jun;125(6):1550-3. doi: 10.1016/s0022-5223(03)00045-x. No abstract available. PMID 12830086
- [Background] Usui A, Ueda Y, Watanabe T, Kawaguchi O, Ohara Y, Takagi Y, Tajima K, Nishikimi N, Ishiguchi T. Clinical results of implantation of an endovascular covered stent-graft via midsternotomy for distal aortic arch aneurysm. Cardiovasc Surg. 2000 Dec;8(7):545-9. doi: 10.1016/s0967-2109(00)00066-1. PMID 11068215
- [Background] Karck M, Kamiya H. Progress of the treatment for extended aortic aneurysms; is the frozen elephant trunk technique the next standard in the treatment of complex aortic disease including the arch? Eur J Cardiothorac Surg. 2008 Jun;33(6):1007-13. doi: 10.1016/j.ejcts.2008.02.030. Epub 2008 Apr 10. PMID 18406159
- [Background] Shrestha M, Pichlmaier M, Martens A, Hagl C, Khaladj N, Haverich A. Total aortic arch replacement with a novel four-branched frozen elephant trunk graft: first-in-man results. Eur J Cardiothorac Surg. 2013 Feb;43(2):406-10. doi: 10.1093/ejcts/ezs296. Epub 2012 May 31. PMID 22653445
- [Background] Patel AY, Eagle KA, Vaishnava P. Acute type B aortic dissection: insights from the International Registry of Acute Aortic Dissection. Ann Cardiothorac Surg. 2014 Jul;3(4):368-74. doi: 10.3978/j.issn.2225-319X.2014.07.06. PMID 25133099
- [Background] Tsai TT, Trimarchi S, Nienaber CA. Acute aortic dissection: perspectives from the International Registry of Acute Aortic Dissection (IRAD). Eur J Vasc Endovasc Surg. 2009 Feb;37(2):149-59. doi: 10.1016/j.ejvs.2008.11.032. Epub 2008 Dec 20. PMID 19097813
- [Background] Jakob H, Tsagakis K. International E-vita open registry. Ann Cardiothorac Surg. 2013 May;2(3):296-9. doi: 10.3978/j.issn.2225-319X.2013.03.10. PMID 23977597